CLINICAL TRIAL: NCT06184399
Title: Efficacy, Safety and Acceptability of Ascending Doses of Ivermectin in Combination With Albendazole for Trichuris Trichiura Infections in Preschool-aged Children: a Single-blind Randomised Controlled Dose-ranging Trial
Brief Title: Efficacy, Safety and Acceptability of Ivermectin ODT in PSAC
Acronym: Iverped
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Iverped_1
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Trichuriasis; Ascariasis; Hookworm Infections
Keywords: Ivermectin; Albendazole; Anthelminthics; Trichuris trichiura; Ascaris lumbricoides; Hookworm; Whipworm; Soil-transmitted helminths
MeSH Terms: conditions — Trichuriasis; Ascariasis; Hookworm Infections; Ancylostomiasis | interventions — Ivermectin; Albendazole; Tablets

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) Treatment allocation will be masked using appearance-matched placebos.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm A: Ivermectin ODT Placebo & Albendazole (Placebo Comparator): Placebo for ivermectin (oro-dispersible tablets) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Albendazole 400 mg Oral Tablet; Drug: Placebo Ivermectin ODT
- Arm B: Ivermectin ODT 100 µg/kg & Albendazole (Experimental): Combination therapy of ivermectin (100 µg/kg using oro-dispersible tablets of 1.5 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Ivermectin 1.5 mg ODT; Drug: Albendazole 400 mg Oral Tablet
- Arm C: Ivermectin ODT 200 µg/kg & Albendazole (Experimental): Combination therapy of ivermectin (200 µg/kg using oro-dispersible tablets of 1.5 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Ivermectin 1.5 mg ODT; Drug: Albendazole 400 mg Oral Tablet
- Arm D: Ivermectin ODT 300 µg/kg & Albendazole (Experimental): Combination therapy of ivermectin (300 µg/kg using oro-dispersible tablets of 1.5 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Ivermectin 1.5 mg ODT; Drug: Albendazole 400 mg Oral Tablet
- Arm E: Ivermectin ODT 400 µg/kg & Albendazole (Experimental): Combination therapy of ivermectin (400 µg/kg using oro-dispersible tablets of 1.5 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Ivermectin 1.5 mg ODT; Drug: Albendazole 400 mg Oral Tablet
- Arm F: Ivermectin standard tablets & Albendazole (Active Comparator): Combination therapy of ivermectin (Stromectol®, 200 µg/kg using tablets of 3 mg) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Interventions: Drug: Ivermectin 3 mg Oral Tablet; Drug: Albendazole 400 mg Oral Tablet

INTERVENTIONS:
Drug: Ivermectin 1.5 mg ODT — Oro-dispersible tablets of 1.5 mg ivermectin
  Arms: Arm B: Ivermectin ODT 100 µg/kg & Albendazole; Arm C: Ivermectin ODT 200 µg/kg & Albendazole; Arm D: Ivermectin ODT 300 µg/kg & Albendazole; Arm E: Ivermectin ODT 400 µg/kg & Albendazole
Drug: Ivermectin 3 mg Oral Tablet — Tablets of 3 mg ivermectin
  Other Names: Stromectol®
  Arms: Arm F: Ivermectin standard tablets & Albendazole
Drug: Albendazole 400 mg Oral Tablet — Tablets of 400 mg albendazole
  Other Names: Zentel®
Drug: Placebo Ivermectin ODT — Placebo for ivermectin ODT
  Arms: Arm A: Ivermectin ODT Placebo & Albendazole

SUMMARY:
This study is a single-blind randomized controlled dose-ranging trial aiming at providing evidence on the on the optimal dose of co-administered ivermectin and albendazole in terms of efficacy, safety and acceptability in preschool-aged children (PSAC; aged 2-5 years) infected with whipworm (Trichuris trichiura) on Pemba Island, Tanzania. Additionally, the pharmacokinetics of the newly developed oro-dispersible tablets (ODTs) and the standard ivermectin tablets (Stromectol®) will be compared in this age group.

As measure of efficacy of the treatment the cure rate (percentage of egg-positive participants at baseline who become egg-negative after treatment) will be determined 14-21 days post-treatment.

DETAILED DESCRIPTION:
This study is a single-blind randomized controlled dose-ranging trial aiming at providing evidence on the optimal dose of co-administered ivermectin and albendazole in terms of efficacy, safety and acceptability in preschool-aged children (PSAC; aged 2-5 years) infected with whipworm (Trichuris trichiura) on Pemba Island, Tanzania. Additionally, the pharmacokinetics of the newly developed ODTs and the standard ivermectin tablets (Stromectol®) will be compared in this age group.

The primary objective of the trial is to comparatively assess the efficacy in terms of cure rate (CR) against T. trichiura infections among PSAC receiving different doses of ivermectin.

The secondary objectives of the trial are to compare the egg reduction rates (ERRs) of the treatment regimens against T. trichiura, to determine the CRs and ERRs of the drugs in study participants co-infected with A. lumbricoides and hookworm, and to evaluate the safety and tolerability of the treatment regimens.

In addition, this study aims to characterize population pharmacokinetics of the ivermectin ODTs compared to standard tablets in T. trichiura infected individuals, and to assess the acceptability of the treatments.

After obtaining informed consent from parents and/or caregivers, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician before treatment. Enrollment will be based on two stool samples, which will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days. All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians.

Randomization of participants into the six treatment arms will be stratified according to intensity of infection and age. All participants will be interviewed before treatment, and at 3 and 24 hours and 14-21 days after treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days post-treatment by collecting another two stool samples.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment. Differences among CRs between treatment arms will be analysed using crude and adjusted logistic regression modeling (adjustment for age, sex and weight). Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs.Using the DoseFinding package of the statistical software environment R, Emax models will be implemented to predict the dose-response curves based on CRs and ERRs.

Adverse events will be compiled into frequency tables and compared between treatment groups using descriptive summary statistics.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 2-5 years (24-71 months; confirmed by birth certificate or similar document)
* having given written informed consent signed by parents/caregivers
* being able and willing to provide two stool samples at baseline and at follow-up assessment (14-21 days)
* having at least two out of four Kato-Katz slides positive for T. trichiura at baseline
* being able and willing to be examined by a study physician before and after treatment

Exclusion Criteria:

* presence or signs of major systemic illness, e.g. fever (temporal body temperature of >38.0°C), severe anaemia (haemoglobin level of <70 g/l)
* history of severe acute disease or unmanaged, severe chronic disease (i.e., condition is not as therapeutically controlled as necessary)
* use of anthelminthic drugs during study period
* known allergy to study medication (i.e., ivermectin or albendazole)
* being prescribed or taking concomitantly medication with known contraindications or drug interactions with the study medication
* concurrent participation in other clinical trials

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Tanzania

REFERENCES:
- [Derived] Sprecher VP, Schnoz A, Biendl S, Hussein HS, Najim SO, Ali MN, Mohammed IS, Ali SM, Hattendorf J, Keiser J. Efficacy and safety of ascending doses of orodispersible ivermectin co-administered with albendazole for Trichuris trichiura infections in preschool-aged children in Tanzania: a single-blind, randomised, controlled, dose-ranging, phase 2 trial. Lancet Infect Dis. 2025 Sep 17:S1473-3099(25)00472-4. doi: 10.1016/S1473-3099(25)00472-4. Online ahead of print. PMID 40975108

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Ivermectin ODT Placebo & Albendazole: Placebo for ivermectin (oro-dispersible tablets, ODT) and albendazole (Zentel®, 1 tablet of 400 mg) administered orally at day 0
  Albendazole 400 mg Oral Tablet: Tablets of 400 mg albendazole
  Placebo Ivermectin ODT: Placebo for ivermectin ODT
Period: Overall Study
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Started | 43 | 44 | 42 | 44 | 44 | 43
Completed | 40 | 42 | 42 | 39 | 40 | 42
Not Completed | 3 | 2 | 0 | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole | Total
Number analyzed (Participants) | 43 | 44 | 42 | 44 | 44 | 43 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (1.1) | 3.6 (1.1) | 3.5 (1.0) | 3.6 (1.0) | 3.5 (1.0) | 3.7 (1.2) | 3.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 24 | 24 | 21 | 26 | 137
  Male | 21 | 24 | 18 | 20 | 23 | 17 | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Tanzania | 43 | 44 | 42 | 44 | 44 | 43 | 260
Trichuris trichiura infection intensity [Count of Participants; unit: Participants]
  Light (<1000 EPG) | 36 | 36 | 34 | 35 | 36 | 34 | 211
  Moderate (1000-9999 EPG) | 7 | 8 | 7 | 9 | 8 | 9 | 48
  Heavy (>9999 EPG) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascaris lumbricoides co-infection [Count of Participants; unit: Participants] | 10 | 13 | 8 | 7 | 9 | 9 | 56
Hookworm co-infection [Count of Participants; unit: Participants] | 8 | 11 | 8 | 10 | 8 | 7 | 52

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate (CR) Against T. Trichiura
Description: The CR will be calculated as the proportion of participants converting from being egg-positive pre-treatment to egg-negative post-treatment.
Time Frame: 14-21 days post-treatment
Population: Available case population
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 40 | 42 | 42 | 39 | 40 | 42
percentage of participants cured (%) | 17.5 [7.3 to 32.8] | 50.0 [34.2 to 65.8] | 83.3 [68.6 to 93.0] | 84.6 [69.5 to 94.1] | 90.0 [76.3 to 97.2] | 73.8 [58.0 to 86.1]

2. Secondary Outcome: Egg Reduction Rate (ERR) Against T. Trichiura (Geometric Mean ERR)
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days post-treatment
Population: Available case population.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 40 | 42 | 42 | 39 | 40 | 42
percent change in egg counts (%) | 65.5 [30.5 to 83.5] | 97.2 [93.9 to 98.8] | 99.7 [99.2 to 99.9] | 99.7 [99.1 to 99.9] | 99.8 [99.5 to 100.0] | 99.2 [97.9 to 99.8]

3. Secondary Outcome: Egg Reduction Rate (ERR) Against T. Trichiura (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Available case population.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 40 | 42 | 42 | 39 | 40 | 42
percent change in egg counts (%) | 30.2 [-11.0 to 54.2] | 88.3 [79.6 to 94.3] | 98.9 [96.8 to 99.7] | 97.9 [94.4 to 99.6] | 98.3 [95.6 to 99.9] | 79.8 [38.7 to 97.2]

4. Secondary Outcome: Cure Rate (CR) Against A. Lumbricoides
Description: as for outcome 1
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 10 | 13 | 8 | 7 | 7 | 9
percentage of participants cured (%) | 100.0 [69.2 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [66.4 to 100.0]

5. Secondary Outcome: Egg Reduction Rate (ERR) Against A. Lumbricoides (Geometric Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 10 | 13 | 8 | 7 | 7 | 9
percent change in egg counts (%) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

6. Secondary Outcome: Egg Reduction Rate (ERR) Against A. Lumbricoides (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with A. lumbricoides at baseline and providing follow-up data.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 10 | 13 | 8 | 7 | 7 | 9
percent change in egg counts (%) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Cure Rate (CR) Against Hookworm
Description: as for outcome 1
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 8 | 11 | 8 | 10 | 7 | 7
percentage of participants cured (%) | 100.0 [63.1 to 100.0] | 45.5 [16.8 to 76.6] | 62.5 [24.5 to 91.5] | 70.0 [34.8 to 93.3] | 71.4 [29.0 to 96.3] | 57.1 [18.4 to 90.1]

8. Secondary Outcome: Egg Reduction Rate (ERR) Against Hookworm (Geometric Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 8 | 11 | 8 | 10 | 7 | 7
percent change in egg counts (%) | 100.0 [100.0 to 100.0] | 93.1 [78.4 to 98.2] | 97.4 [83.0 to 99.8] | 97.9 [92.4 to 100.0] | 98.6 [94.0 to 100.0] | 97.1 [87.4 to 99.7]

9. Secondary Outcome: Egg Reduction Rate (ERR) Against Hookworm (Arithmetic Mean ERR)
Description: as for outcome 2
Time Frame: 14-21 days post-treatment
Population: Subset of participants co-infected with hookworm at baseline and providing follow-up data.
Measure: Mean (95% Confidence Interval); unit: percent change in egg counts (%)
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 8 | 11 | 8 | 10 | 7 | 7
percent change in egg counts (%) | 100.0 [100.0 to 100.0] | 85.7 [54.4 to 93.1] | 88.9 [66.7 to 99.2] | 92.8 [83.6 to 100.0] | 92.2 [82.8 to 100.0] | 62.3 [38.6 to 98.6]

10. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Participants will be monitored at the site for 3 hours following treatment for any acute AEs and reassessment will be done at 24h post-treatment. In addition, participants will be interviewed 3 and 24 hours after treatment and retrospectively at days 14-21 about the occurrence of AEs.
Time Frame: 3 hours, 24 hours and 14-21 days post-treatment
Population: All participants receiving treatment.
Measure: Number; unit: participants
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
Number analyzed (Participants) | 43 | 44 | 42 | 44 | 44 | 43
participants
  3 hours: Abdominal pain | 1 | 1 | 1 | 0 | 0 | 1
  3 hours: Diarrhoea | 0 | 0 | 0 | 0 | 0 | 0
  3 hours: Vomiting | 0 | 0 | 0 | 0 | 0 | 0
  24 hours: Abdominal pain | 3 | 2 | 0 | 1 | 2 | 0
  24 hours: Diarrhoea | 1 | 0 | 0 | 0 | 4 | 0
  24 hours: Vomiting | 0 | 0 | 0 | 0 | 2 | 0
  14-21 days: Abdominal pain | 0 | 0 | 0 | 0 | 0 | 0
  14-21 days: Diarrhoea | 0 | 0 | 0 | 0 | 0 | 0
  14-21 days: Vomiting | 0 | 0 | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Blood Concentration of Ivermectin
Description: For characterization of population pharmacokinetics (PK), ivermectin concentration will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a lower limit of quantification of 1-5 ng/ml.
Time Frame: 0 to 24 hours post-treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Acceptability of ODT Assessed by Visual Analogue Scale (0-100 mm)
Description: To determine the acceptability of ivermectin ODTs compared to standard tablets, the palatability of each formulation will be rated by children aged 4-5 years using a visual analogue scale with continuous scores from 0 mm (worst taste) to 100 mm (best taste).
Time Frame: 15 min post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2-3 weeks
Arm/Group | Arm A: Ivermectin ODT Placebo & Albendazole | Arm B: Ivermectin ODT 100 µg/kg & Albendazole | Arm C: Ivermectin ODT 200 µg/kg & Albendazole | Arm D: Ivermectin ODT 300 µg/kg & Albendazole | Arm E: Ivermectin ODT 400 µg/kg & Albendazole | Arm F: Ivermectin Standard Tablets & Albendazole
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 0/42 | 0/44 | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/42 | 0/44 | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 4/43 | 3/44 | 1/42 | 1/44 | 7/44 | 1/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ivermectin ODT Placebo & Albendazole (N=43) | Arm B: Ivermectin ODT 100 µg/kg & Albendazole (N=44) | Arm C: Ivermectin ODT 200 µg/kg & Albendazole (N=42) | Arm D: Ivermectin ODT 300 µg/kg & Albendazole (N=44) | Arm E: Ivermectin ODT 400 µg/kg & Albendazole (N=44) | Arm F: Ivermectin Standard Tablets & Albendazole (N=43)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT06184399/Prot_SAP_000.pdf